CLINICAL TRIAL: NCT04000178
Title: COMPARISON OF SILICONE VERSUS POLYURETHANE URETERAL STENTS: A PROSPECTIVE CONTROLLED STUDY
Brief Title: OPTIMAL STENTS DURING RENAL COLIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, nariman.gadjiev, Head of endourology, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217
Record Dates: First submitted 2019-06-23; First posted 2019-06-27 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Ureteral Stent Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Other): patients who received polyurethane stents
  Interventions: Device: polyurethane stent
- group B (Experimental): patients who received silicone stents
  Interventions: Device: silicone stent

INTERVENTIONS:
Device: polyurethane stent — patients were prospectively enrolled in the study and stratified (non-randomly) into either group A - polyurethane - control group or group B - silicone - experimental group
  Arms: group A
Device: silicone stent — silicone stent
  Arms: group B

SUMMARY:
From June 2018 to October 2018, patients from two distinct clinical centers were prospectively enrolled in the study and stratified (non-randomly) into either control group A, patients who received polyurethane stents (Rüsch, Teleflex), or experimental group B, patients who received silicone stents (Cook Medical). Each participant completed a survey one hour after stent insertion, in the middle of the stent dwelling period, and before stent removal or ureteroscopy noting body pain and overactive bladder via the visual analog scale pain (VASP) and overactive bladder (OAB) awareness tool, respectively. Additionally, the successfulness of stent placement, hematuria, number of unplanned visits, and stent encrustation rates were assessed within each group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included age (18 to 60 years old),
* confirmed ureteral stone
* prescribed ureteral stent placement for pain syndrome relief

Exclusion Criteria:

* an active urinary tract infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
body pain | 4 weeks
  At each follow-up appointment, patients completed a survey in which the visual analog scale pain (VASP) was filled
bladder overactivity | 4 weeks
  At each follow-up appointment, patients completed a survey in which the "bladder awareness tool" (VASP) was filled

CONTACTS AND LOCATIONS:
Locations (1):
- First Pavlov Saint Petersburg University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gadzhiev N, Gorelov D, Malkhasyan V, Akopyan G, Harchelava R, Mazurenko D, Kosmala C, Okhunov Z, Petrov S. Comparison of silicone versus polyurethane ureteral stents: a prospective controlled study. BMC Urol. 2020 Feb 3;20(1):10. doi: 10.1186/s12894-020-0577-y. PMID 32013936